CLINICAL TRIAL: NCT04071171
Title: Comparison of Biphozyl® and Phoxilium® as a Replacement Fluid During CVVH for AKI in Adults and Their Effects on pH-, Bicarbonate-levels and Respiratory Situation - A Prospective, Randomized, Controlled, Open, Cross-over, Phase II, Single-center Pilot Study [BiPhox-Trial]
Brief Title: Comparison of Biphozyl® and Phoxilium® as a Replacement Fluid During CVVH for AKI in Adults and Their Effects on pH-, Bicarbonate-levels and Respiratory Situation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No. 2019-001262-15
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Critically Ill; Acute Kidney Injury; Renal Replacement Therapy; Continuous Renal Replacement Therapy; Continuous Veno-Venous Hemofiltration; Replacement Fluid; Phoxilium; Biphozyl; Anticoagulation; Regional Citrate Anticoagulation
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phoxilium® (Active Comparator)
  Interventions: Drug: CVVH with Phoxilium® in the first 48h after randomization; Drug: CVVH with Phoxilium® in the second 48h after randomization (after previous 48h with Biphozyl®)
- Biphozyl® (Experimental)
  Interventions: Drug: CVVH with Biphozyl® in the first 48h after randomization; Drug: CVVH with Biphozyl® in the second 48h after randomization (after previous 48h with Phoxilium®)

INTERVENTIONS:
Drug: CVVH with Phoxilium® in the first 48h after randomization — After randomization into the Phoxilium®-group, CVVH will be initiated with Phoxilium® as a replacement fluid and maintained for 48h, respectively until the crossover. Anticoagulation is delivered as pre-filter RCA with Regiocit® (Gambro Lundia AB, Sweden). For antagonisation of Regiocit®, a calcium solution (calcium chloride, with or without magnesium chloride) will be used post-filter.
  Arms: Phoxilium®
Drug: CVVH with Biphozyl® in the first 48h after randomization — After randomization into the Biphozyl®-group, CVVH will be initiated with Biphozyl® as a replacement fluid and maintained for 48h, respectively until the crossover. Anticoagulation is delivered as pre-filter RCA with Regiocit® (Gambro Lundia AB, Sweden). For antagonisation of Regiocit®, a calcium solution (calcium chloride, with or without magnesium chloride) will be used post-filter.
  Arms: Biphozyl®
Drug: CVVH with Phoxilium® in the second 48h after randomization (after previous 48h with Biphozyl®) — 48h post randomization, respectively after the cross-over CVVH will be continued with Phoxilium® for another 48h. Anticoagulation is delivered as pre-filter RCA with Regiocit® (Gambro Lundia AB, Sweden). For antagonisation of Regiocit®, a calcium solution (calcium chloride, with or without magnesium chloride) will be used post-filter.
  Arms: Phoxilium®
Drug: CVVH with Biphozyl® in the second 48h after randomization (after previous 48h with Phoxilium®) — 48h post randomization, respectively after the cross-over CVVH will be continued with Biphozyl® for another 48h. Anticoagulation is delivered as pre-filter RCA with Regiocit® (Gambro Lundia AB, Sweden). For antagonisation of Regiocit®, a calcium solution (calcium chloride, with or without magnesium chloride) will be used post-filter.
  Arms: Biphozyl®

SUMMARY:
The primary objectives of the BiPhox-Trial are to demonstrate, that the use of Biphozyl® as a replacement fluid in adult critically ill acute kidney injury (AKI) patients, results in a lower rate of pH excursions and of bicarbonate (HCO3-) excursions compared to the use of Phoxilium® during the studied continuous veno-venous hemofiltration (CVVH) interval with regional citrate anticoagulation (RCA).

The secondary objectives of the BiPhox-Trial are to evaluate the time to pH level normalization and the HCO3- substitution rates after initiation of CVVH treatment. Further, to demonstrate that the use of Biphozyl® as a replacement fluid in adult critically ill AKI patients, results in a more stable acid-base-status as well as improved respiratory situation due to lower intracorporeal HCO3- and carbon dioxide levels compared to the use of Phoxilium® during the studied CVVH interval with RCA.

DETAILED DESCRIPTION:
After being fully eligible by meeting all inclusion and none of the exclusion criteria, participants will be randomly assigned to one of two groups, either the Phoxilium® - Group or Biphozyl® - Group. After randomization, patients receive either Phoxilium® or Biphozyl® for CVVH initiation and maintenance as a replacement fluid during the first 48 hours (h) of treatment. After the first 48h of CVVH with either Phoxilium® or Biphozyl® a cross-over follows, with another 48h of CVVH with the opposite replacement fluid (Phoxilium® switched to Biphozyl® or Biphozyl® switched to Phoxilium®). In comparison, all patients should receive one session of CVVH with 96h. Resulting from 48h of CVVH with Phoxilium® and 48h of CVVH with Biphozyl® as a replacement fluid. The order is determined by randomization.

Anticoagulation is always delivered as pre-filter RCA with Regiocit® (Gambro Lundia AB, Sweden). For antagonisation of Regiocit®, a calcium solution (calcium chloride, with or without magnesium chloride) will be used post-filter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admission to Intensive Care Unit
3. Indication for CVVH as determined by the attending physician
4. Planned CVVH treatment time ≥ 48 hours
5. Written informed consent or deferred consent or legally acceptable representative consent

Exclusion Criteria:

1. Lack of commitment to provide CVVH as part of limitation of ongoing life support
2. Presence of a drug overdose that may result in acid-base-disorders and/or a shift of electrolytes
3. Receipt of CVVH within the previous 72 hours
4. Dialysis dependent end-stage renal disease
5. Pregnancy, must be ruled out by anamnesis and/or blood or urine pregnancy test
6. Combination of severely impaired liver function and shock with muscle hypoperfusion
7. Co-enrollment in another trial, which could have a plausible interaction with the acid-base-status and/or any electrolytes
8. Subjects, who are legally exempted from participation in clinical trials (e.g. persons held in an institution by legal or official order)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
pH | 96 hours (48h of CVVH with Phoxilium® vs. 48h of CVVH with Biphozyl®)
  Rate of pH excursions from a set range of 7.35-7.45.
HCO3- | 96 hours (48h of CVVH with Phoxilium® vs. 48h of CVVH with Biphozyl®)
  Rate of HCO3- excursions from a set range of 22-26 mmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joannidis, Univ.-Prof., MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Division of Intensive Care and Emergency Medicine, Department of Internal Medicine, Medical University Innsbruck, Anichstrasse 35, 6020, Innsbruck, Austria, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Perschinka F, Koglberger P, Kohler A, Lehner GF, Peer A, Maier S, Ulmer H, Bellmann R, Forni LG, Joannidis M. Comparison of two different bicarbonate replacement fluids during CVVH with RCA: a prospective, randomized, controlled trial. Intensive Care Med. 2025 Dec;51(12):2354-2366. doi: 10.1007/s00134-025-08175-7. Epub 2025 Nov 17. PMID 41247497
- [Derived] Koglberger P, Perschinka F, Klein SJ, Mayerhofer T, Maier S, Ulmer H, Bellmann R, Joannidis M. Protocol of the Comparison of Two Different Bicarbonate Replacement Fluids during Continuous Veno-Venous Hemofiltration with Regional Citrate Anticoagulation: A Prospective, Randomized, Controlled Trial. Blood Purif. 2025;54(12):723-732. doi: 10.1159/000547401. Epub 2025 Aug 4. PMID 40759107